CLINICAL TRIAL: NCT00914043
Title: Biobehavioral Mechanisms of Fatigue in Patients Treated on NSABP B-45: A Phase III Clinical Trial Comparing Adjuvant Sunitinib Malate to Placebo in Women With Residual Invasive Breast Cancer Following Neoadjuvant Chemotherapy
Brief Title: Studying Biological Markers of Fatigue in Women With Residual Invasive Breast Cancer Enrolled on Clinical Trial NSABP-B-45
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn as NCI rescinded approval for parent study NSABP-B-45
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NSABP B-45.1; NSABP-B-45.1
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer; Fatigue
Keywords: fatigue; HER2-negative breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Gene Expression Profiling; Microarray Analysis; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Reverse Transcriptase Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay; Therapeutics

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: biologic sample preservation procedure
Other: enzyme-linked immunosorbent assay
Other: laboratory biomarker analysis
Procedure: fatigue assessment and management

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to fatigue.

PURPOSE: This research study is looking at biological markers of fatigue in women with residual invasive breast cancer enrolled on clinical trial NSABP-B-45.

DETAILED DESCRIPTION:
OBJECTIVES:

* To collect serial blood specimens at each time point that quality of life and patient-reported outcome assessments are performed in women with residual invasive breast cancer concurrently enrolled on and participating in the Behavioral and Health Outcomes component of clinical trial NSABP-B-45.
* To prepare, separate, and store the blood specimens at the NSABP Serum Bank at Baylor College of Medicine Breast Center into components for future DNA, RNA, and plasma analysis.
* To analyze specific proinflammatory cytokines, genetic polymorphisms, and RNA expression arrays in collaborating laboratories at University of California, Los Angeles (UCLA).
* To examine the association between markers of inflammation and symptoms of fatigue among patients treated with sunitinib malate or placebo on clinical trial NSABP-B-45.
* To examine the relationship between single-nucleotide polymorphisms in the promoter regions of IL-1 and IL-6 and symptoms of fatigue in these patients.
* To examine the relationship between RNA expression profiles and fatigue and compare the pattern of expression in these patients.

OUTLINE: This is a multicenter study.

Patients undergo blood sample collection* at baseline and then at 3, 6, 12, 18, and 24 months for analysis of plasma concentrations of inflammatory biomarkers (IL-1ra, sTNFRII, sIL-6R, and C-reactive protein) by ELISA; DNA polymorphisms in the promoter regions of IL-6 and IL-1 by TaqMan PCR; and RNA gene expression signaling pathways by RT-PCR assays and microarray.

NOTE: *Blood samples are collected at the same time points that the Behavioral and Health Outcomes quality of life and patient-reported outcomes questionnaires are completed on clinical trial NSABP-B-45.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of residual invasive breast cancer

  * Stage II, IIIA, or IIIB disease
  * HER2/neu-negative disease
* Randomized to receive either sunitinib malate or placebo on clinical trial NSABP-B-45

  * Has not started therapy on clinical trial NSABP-B-45
* Has completed baseline Behavioral and Health Outcome questionnaires on clinical trial NSABP-B-45
* Hormone-receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Biological and behavioral predictors of fatigue in breast cancer patients at 12 and 24 months after randomization and initiation of treatment on clinical trial NSABP-B-45
Relationship between specific single-nucleotide polymorphisms in the promoter regions of IL-1 and IL-6 and circulating markers of inflammation and symptoms of fatigue
Relationship between RNA gene expression pathways and symptoms of fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc